CLINICAL TRIAL: NCT04432961
Title: A Database and Analytics Study of Free Text Clinical Notes and Structured Data to Investigate Phenotype Associations With Outcomes in Patients With COVID-19
Brief Title: Natural Language Processing (NLP) Analysis of Free Text Notes to Investigate Coronavirus (COVID-19)
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr Sapna Trivedi, Doctor, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A095625
Record Dates: First submitted 2020-06-15; First posted 2020-06-16 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
Keywords: Natural Language Processing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective cohort study investigating clinical notes using Natural Language Processing in combination with structured data from the Electronic Health Record (EHR) to create a database for analytics to identify features associated with outcomes.

DETAILED DESCRIPTION:
Patients admitted to Cambridge University Hospitals (CUH)with COVID-19 have undergone routine clinical documentation and specific investigation and testing for COVID-19. The pathway for these patients ranges from supportive measures on the ward to deterioration requiring Intensive therapy Unit (ITU) admission and ventilatory support. Patients are also at risk of developing complications such as Acute Kidney Injury and thromboembolism. Identification of the risk factors for these and other outcomes such as the requirement for ventilation remain a challenge and reviewing the clinical data for these patients is critical in the understanding of the relationship between patient characteristics and outcomes.

There is data available in structured fields in the EHR, however, this is sometimes incomplete and inaccurate. An assessment of the free text clinical notes provides an opportunity to fill in the gaps and provide a much richer dataset for evaluation. We plan to use Natural Language Processing (NLP) (a field of machine learning that allows computers to analyse human language) to review Discharge Summaries of patients admitted to hospital with COVID-19 and convert free text data into structured data for analysis.

The NLP techniques developed by Dr Collier's team include methods for coding of free texts to SNOMED CT and other biomedical ontologies. These methods, based on statistical machine learning from human annotated texts, have been benchmarked for scientific texts and social media. In this project we intend to adapt these techniques for patient records. The techniques will require a number of human annotated patient records in order to adapt. The NLP output will be combined with structured data from the EHR and undergo statistical analysis to identify the rates of complications in patients with COVID-19 and risk factors associated with these. This may help to guide management decisions by earlier intervention to prevent poor outcomes in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age range: 18 to 100 years
* Patients admitted to Cambridge University Hospitals with confirmed COVID-19 on lab testing

Exclusion Criteria:

Children and patients with a negative COVID test.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Cambridge University Hospitals NHS Foundation Trust with confirmed COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
research database of EHR records from COVID-19 patients processed using NLP tools for named entity recognition and linking adapted to CUH EMR data to identify variables of interest | 1 year
  Our overarching hypothesis is that the NLP-extracted data from the free-text discharge summary can be combined with structured data from the EMR to yield insights into the development of complications. Patient with severe disease requiring ITU admission and non severe disease managed on an inpatient ward will be included. The variables of interest will include patient characteristics and specific encounter related information including length of stay and baseline investigations (e.g., blood tests) and interventions received

SECONDARY OUTCOMES:
A set of annotation guidelines to produce human-expert (gold) labelled data for a subset of the EHR | 6 months
A comparison of the NLP output to terms in the structured problem list to identify missing terms in the structured problem list | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University NHS Foundation Trust, Cambridge, United Kingdom